CLINICAL TRIAL: NCT03283865
Title: Does Use of Ultrasound Reduce the Rate of Sham Caudal Block in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: doesnt meet criteria for clinical trial reporting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-40844
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Regional Anesthesia Morbidity

STUDY DESIGN:
Intervention Model Description: Single blinded prospective trial in which all patients serve as their own clinical control group.
Masking Description: Single blinded prospective trial in which all patients serve as their own clinical control group.
  Provider doing the procedure will be blinded to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ultrasound (Experimental): The attending anesthesiologist will perform or instruct the placement of a caudal block according to their standard of practice. At the time of administration of local anesthetic into the caudal space, the study collaborator (SC) will ultrasound the caudal space keeping the provider placing the block blinded to the imaging. The provider placing the block will inject 0.5mL of saline. The provider will then be asked to state if they are correctly in the caudal space or not. If the provider feels they are not in the caudal space, they will re-do the procedure. If the provider fails to identify incorrect location and this is noted by ultrasound, the SC will inform the provider to re-do the procedure.
  All study participants will have ultrasound used for caudal block.
  Interventions: Diagnostic Test: Ultrasound guidance for caudal block

INTERVENTIONS:
Diagnostic Test: Ultrasound guidance for caudal block — The attending anesthesiologist will perform or instruct the placement of a caudal block according to their standard of practice. At the time of administration of local anesthetic into the caudal space, the study collaborator (SC) will ultrasound the caudal space keeping the provider placing the block blinded to the imaging. The provider placing the block will inject 0.5mL of preservative free saline. The provider will then be asked to state if they are correctly in the caudal space or not. If the provider feels they are not in the caudal space, they will re-do the procedure. If the provider fails to identify incorrect location and this is noted by ultrasound, the SC will inform the provider to re-do the procedure

SUMMARY:
Caudal blocks are one of the most commonly performed regional anesthetics in children and are performed daily for a host of infra-umbilical surgical procedures. A caudal block is an epidural injection, most commonly of local anesthetic into the epidural space as accessed via the sacral hiatus. In children, the sacral hiatus is a normally occurring aperture in which the epidural space may be accessed with extremely minimal risk; as neural tissue ends more proximally. Due to this measure of safety, caudal blocks are preferred in children when compared with standard lumbar epidurals. Caudal blocks are performed blindly using palpation and tactile feedback to assess if the medication is being administered in the correct location. As a result of blind injection, administration of local anesthetic totally or partially outside of the correct site can often be unnoticed or identified after a significant volume has already been injected. With the potential for toxicity of local anesthetic, this may result in either the inability to give a complete dose or an unintentional and often unnoticed sham block "incorrect site of injection".

DETAILED DESCRIPTION:
Caudal blocks are one of the most commonly performed regional anesthetics in children and are performed daily for a host of infra-umbilical surgical procedures. A caudal block is an epidural injection, most commonly of local anesthetic into the epidural space as accessed via the sacral hiatus. In children, the sacral hiatus is a normally occurring aperture in which the epidural space may be accessed with extremely minimal risk; as neural tissue ends more proximally. Due to this measure of safety, caudal blocks are preferred in children when compared with standard lumbar epidurals. Caudal blocks are performed blindly using palpation and tactile feedback to assess if the medication is being administered in the correct location. As a result of blind injection, administration of local anesthetic totally or partially outside of the correct site can often be unnoticed or identified after a significant volume has already been injected. With the potential for toxicity of local anesthetic, this may result in either the inability to give a complete dose or an unintentional and often unnoticed sham block "incorrect site of injection".

Use of ultrasound has been proposed for identification of caudal block placement and correct medication spread. However, a recent review of the Pediatric Regional Anesthesia Network database reveals that ultrasound is reportedly only used in less that 3% of blocks. The benefit of ultrasound is safe and real-time confirmation of injection. Ultrasound allows the provider to determine with minimal local anesthetic or even saline injection if the correct space is accessed. Without ultrasound, failed blocks are either identified after significant percentage of the total dose of local anesthetic is incorrectly administered or intra or post operatively when the patient demonstrates a significant opioid requirement. This is problematic given that one of the primary benefits of a caudal block in children is the ability to avoid opioids.

Review of local practice here at Texas Children's Hospital for quality improvement purposes revealed a failure rate of caudal blocks to be 18%. Failure was defined as a heart rate increase with incision of >20% despite a caudal block and >1MAC of gas for the patient age. These patients all required opioids both intra and post operatively in addition to surgical levels of inhaled anesthetic agent.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 0-84 months
* Infra-umbilical procedure for which a caudal block is already planned
* American Society of Anesthesiology classifications of 1,2 or 3

Exclusion Criteria:

* Incarcerated hernias
* Emergency procedures
* Local Anesthetic allergy
* Sacral dimple
* Rash over sacrum
* Parents/legal guardians unable to consent for surgical procedure in English language Foster Care/Child protective services as guardians
* Parental Refusal for caudal block or study participation
* American Society of Anesthesiology classifications other than 1,2 or 3

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Identify the rate at which blindly placed caudal blocks are not within the epidural space | 15 minutes
  Assess the percentage of providers not recognizing wrong site of injection without ultrasound

SECONDARY OUTCOMES:
Identify the rate at which ultrasound can guide a wrong block into the correct location | 15 minutes
  Assess the number of blocks that are require the use of ultrasound to redirect needle into caudal space
Identify if lack of heart rate change on incision can predict successful placement when medication administration is successfully confirmed with ultrasound | 15 minutes
  With ultrasound identification of correct caudal injection, (successful block), does lack of heart rate change correlated with successful block
Identify if after using ultrasound to visualize placement, if concentrations of inhaled agents may be reduced in children | 30 minutes to 3 hours
  With demonstration of successful caudal injection, can inhaled agent concentration be reduced as calculated by MAC hours

CONTACTS AND LOCATIONS:
Overall Officials: Adam C Adler, MD, FAAP, Principal Investigator — Texas Childrens Hospital
Locations (1):
- Texas childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03283865/Prot_SAP_000.pdf